CLINICAL TRIAL: NCT01788410
Title: MRI-Guided Cryoablation of Head, Neck and Spine Nerves and Facets Using the Advanced Multimodality Image Guided Operating(AMIGO) Suite
Brief Title: MRI-Guided Cryoablation to Alleviate Pain in Head, Neck and Spine
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Thomas C. Lee, MD, Brigham and Women's Hospital
Other Study IDs: 2012-P-002071
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Facet Joints; Degeneration; Neuropathy; Neuralgia
Keywords: Cryoablation; Nerves; Facet joint; Pain; Neuralgia; Neuropathy; Image-guided
MeSH Terms: conditions — Neuralgia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cryoablation under image guidance: Patients with facet joint disease, or compressed or damaged nerve roots causing pain in the head, neck or spine. Procedures performed with MRI Seednet Cryotherapy System (Galil Medical).
  Interventions: Procedure: Cryoablation under image guidance; Device: MRI Seednet Cryotherapy System (Galil Medical)

INTERVENTIONS:
Procedure: Cryoablation under image guidance — Observing efficacy of cryoablation to nerves and facet joints for the treatment of radicular pain and pain resulting from facet joint disease.
  Other Names: MRI Seed Net Cryotherapy Unit (Galil Medical); Siemens IMRIS
Device: MRI Seednet Cryotherapy System (Galil Medical) — Observing efficacy of cryoablation to nerves and facet joints for the treatment of radicular pain and pain resulting from facet joint disease.
  Other Names: FDA Approved; Cryoablation under image guidance

SUMMARY:
The objective of this study is to provide pain relief to patients with facet joint disease or head and neck pain related to compression of a nerve root. The goal is to provide palliative care with superior efficacy and longer relief compared to current methods.

DETAILED DESCRIPTION:
Nerve ablation is used therapeutically to produce temporary anesthesia and diagnostically to locate the source of pain. Ablation, or purposeful destruction of tissue, relieves facet joint pain and pain related to nerve damage by disabling pain-transmitting nerves. Cryoablation for pain management is particularly useful when other modalities are too difficult to perform or have a high incidence for complications or side effects.

Currently nerve ablation is performed with bupivacaine and alcohol, but MRI-guided cryoablation of nerves and facets may result in superior efficacy and longer relief. Cryotherapy techniques provide long term analgesia and help alleviate intractable pain for patients with facet joint pain and neuralgia.

Minimally invasive Magnetic Resonance (MR)-guided ablation of nerves and facets may lead to decreased procedure time and increased relief of pain due to cancer or nerve degeneration. With the advent of the Advanced Multimodality Image Guided Operating Suite (AMIGO) at the Brigham and Women's Hospital, we have exceptional capabilities for minimally invasive image-guided procedures, including different ablation techniques. The AMIGO suite is equipped with hardware that will keep the patient stationary while the Magnetic Resonance Imaging scanner moves to the patient. Additionally, the monitoring software within the AMIGO suite allows clinicians to instantaneously analyze the imaging information which significantly reduces the risk of injury to adjacent structures.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be willing and able to sign a written informed consent document.
* Patients must have facet joint disease or pain due to a damaged or compressed nerve that would benefit from a minimally invasive image-guided procedure (i.e., adjacent to critical structures, better visualized under 3 Tesla MRI than CT)
* Subjects must be able to adhere to the visit schedules and attend pre and post imaging.
* Participants must be at least 18 years of age
* Participants must have an estimated life expectancy of >8 weeks in the opinion of the clinician.

  * Patients with radiculopathy must have the cause of pain confirmed by a nerve block within 3 months prior to ablation

Exclusion Criteria:

* Contraindications to MRI and Gadolinium- (i.e. estimated Glomerular Filtration Rate <60ml/min, metal clips)
* Pregnant or breastfeeding woman are excluded from this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects must be 18 years of age and will be selected among patients who have a pain related to facet joint disease, nerve degeneration or compression. Subjects must benefit from a minimally invasive treatment option.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Eliminating radicular pain or pain caused by spinal disease. | 1 month
  We will be grading patients pain using the "Brief Pain Inventory" pre-ablation and 1 month post-ablation.

SECONDARY OUTCOMES:
Long term radicular pain relief | 1 year
  We are attempting to produce long-term pain relief through cryoablation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Lee, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Brigham and Women's Hospital Tumor Ablation Program — http://www.brighamandwomens.org/Departments_and_Services/radiology/services/abdominalimaging/TumorAblationProgram.aspx
- See also: AMIGO Operating Suite, Brigham and Women's Hospital (BWH) — https://ncigt.org/